CLINICAL TRIAL: NCT00386438
Title: Efficacy of Honan Balloon in Intraocular Pressure Reduction Before Phacoemulsification
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 391/47
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-10

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

INTERVENTIONS:
Procedure: Honan balloon application

SUMMARY:
-Does Honan balloon reduce intraocular pressure preoperatively?

DETAILED DESCRIPTION:
-Does Honan balloon improve surgeon's satisfaction and patients' pain score when compared to no honan group?

ELIGIBILITY:
Inclusion Criteria:

* cataract patient,who plan to undergo phacoemulsification
* no previous ocular surgery

Exclusion Criteria:

* one eye
* high myopia
* Use ASA or anticoagulants
* History of glaucoma or ocular hypertension
* uncooperative patients

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-12; Study Completion 2006-07

PRIMARY OUTCOMES:
intraocular pressure reduction

SECONDARY OUTCOMES:
pain score

CONTACTS AND LOCATIONS:
Overall Officials: Thitima Lunchakonsiripan, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial hospital, Patumwan, Bangkok, Thailand

REFERENCES:
- See also: Faculty of Medicine,Chulalongkorn University — http://www.md.chula.ac.th